CLINICAL TRIAL: NCT00244192
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Effects of Infliximab (Remicade) on Fat Free Mass in Patients With Moderate to Severe COPD Suffering From Cachexia
Brief Title: Effects of Infliximab (Remicade) on Fat Free Mass in Patients With Moderate to Severe COPD Suffering From Cachexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Integrated Rehabilitation and Organ Failure Horn (Other)
Collaborators: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EU-073
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2005-10

CONDITIONS: COPD; Cachexia
Keywords: COPD; infliximab; Remicade; inflammation; cachexia; fat-free mass; health status; exercise capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cachexia; Inflammation | interventions — Infliximab

INTERVENTIONS:
Drug: infliximab (Remicade)

SUMMARY:
The purpose of this study is to determine whether infliximab is effective on fat-free mass in the treatment of patients with moderate to severe COPD suffering from cachexia.

DETAILED DESCRIPTION:
COPD is a multicomponent disease characterized by abnormal inflammatory response of the lungs to noxious particles that accompanied by systemic effects like weight loss, muscle wasting, reduced functional capacity and health status. A persistent systemic inflammatory response reflected by enhanced levels of acute phase proteins like C-reactive protein (CRP) or pro-inflammatory cytokines such as tumor necrosis factor (TNF) - α, is present in COPD. There are several studies that indicate that an increased systemic inflammator response is associated with weight loss, cachexia (loss of fat-free muscle mass), physical functioning and health status.

Cachexia associated with systemivc inflammation can not always readily be overcome by nutritional intervention alone.

The hypothesis of this study is that infliximab therapy (3 infusions with 5 mg/kg infliximab or placebo 1:1 on week 0, 2 and 6) will increase fat-free mass relatively to placebo by decreasing inflammation. Secondary endpoints are: lung function, muscle function, exercise capacity and health status. On week 8, 12 and 26 follow-up measurements will be done.

ELIGIBILITY:
Inclusion Criteria:

1. COPD acording GOLD with FEV1/FVC ratio < 70%, and post-bronchodilator FEV1 > 20% but < 80% of predicted and an FEV1 of >500ml.

2. Fat Free Mass Index : <17.5 kg/m2 in males, <15 kg/m2 in females. 3. Symptomatic (eg, chronic cough, sputum production, shortness of breath) for at least 2 months 4. >= 40 years of age and ≤ 80 years of age 5. History of >=10 pack years of smoking 6. Men and women of childbearing potential must use adequate birth control measures at least one month prior to screening and for the duration of the study and should continue such precautions for 6 months after receiving the last infusion.

7. Ability to adhere to the study visit schedule and other protocol requirements 8. Provide signed, written informed consent prior to participation in the study 9. Be adequately immunized against S. pneumoniae. Patients enrolling in the study in autumn and winter months should be immunized against influenza 10. The screening laboratory test results must meet the following criteria:

1. Hemoglobin >= 8.5 g/dL
2. WBC >= 3.5 x 109/L
3. Neutrophils >= 1.5 x 109/L
4. Platelets >= 100 x 109/L
5. SGOT (AST) and alkaline phosphatase levels must be within 3 times the upper limit of normal range for the laboratory conducting the test.
6. TSH within the normal range of 0.3 to 5 mIU/L. 11. Are considered eligible according to the tuberculosis (TB) eligibility assessment, screening, and early detection of reactivation rules

   Exclusion Criteria:
   1. > 11% increase in FEV1 as % of predicted after a fixed dose of bronchodilator (200 µg inhaled salbutamol)
   2. >12% variation between screening and baseline FEV1 assessments
   3. FEV1 < 500 ml
   4. Patients with asthma as main component of their obstructive airways disease
   5. Moderate or severe exacerbation of COPD within previous 2 months
   6. History or clinical signs of severe cor pulmonale, or pulmonary hypertension, severe right or left sided cardiac failure, serious arrhythmias, myocardial infarction or cardiac interventions within 6 months of screening.

   Exclusion criteria on echocardiogram:

   Exclude patients with right-sided heart defects, as defined by any 1 of the following 3 echocardiography criteria:
   1. Right ventricular size increased, with an inlet diameter of >5cm
   2. Moderate-to-severe tricuspid valve regurgitation
   3. Right ventricular (RV)-right atrial (RA) pressure drop of >50 mmHg Exclusion of patients with left ventricular ejection fraction (LV EF) of <40%, as measured on echocardiography.

   Exclusion criteria on electrocardiogram:

   Exclude patients with the following arrhythmias identified on electrocardiography (ECG):
   1. Fast atrial fibrillation at ventricular rate of >90/min
   2. Atrial-ventricular conduction delay of grade 2 or higher : excludes 2nd and 3rd degree heart block.
   3. Left bundle branch block, with QRS complex >120msec.
   4. Ventricular arrhythmias: ventricular tachycardia and trigeminy.

   7. Chronic respiratory failure (PaO2 < 7.3kPa with or without hypercapnia) and patients requiring long term oxygen therapy.

   8. Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to screening or planned participation in pulmonary rehabilitation during the study 9. Stopping smoking or attending a smoking cessation class within 6 weeks of enrollment.

   10. Known a1 antitrypsin deficiency 11. Serious acute infections (eg, hepatitis, pneumonia or pyelonephritis) in the previous 3 months 12. Major surgery in the previous 3 months 13. Women who are pregnant, nursing, or planning pregnancy within one year after screening (i.e., approximately 6 months following last infusion) 14. Use of any investigational drug within 1 month prior to screening or within 5 half?lives of the investigational agent, whichever is longer 15. Treatment with any other therapeutic agent targeted at reducing TNFa (e.g. pentoxifylline, thalidomide, etanercept, etc.) within 3 months of screening. Treatment with immunosuppressive or cytotoxic therapy.

   16. Previous administration of infliximab 17. Known allergy to murine products 18. Are considered ineligible according to the TB eligibility assessment, screening, and early detection of reactivation rules defined in Section 4.3.

   19. Have or have had an opportunistic infection (eg, herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.

   20. Have a chest radiograph at screening that shows evidence of malignancy, infection, or any abnormalities suggestive of TB 21. Have had an opportunistic infection (e.g. herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months of screening.

   22. Documented HIV infection. 23. Positive serology for active hepatitis B or C based on all subjects being tested at screening. A positive result will indicate referral to a consultant Hepatologist for further investigation and support.

   24. Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, cardiac, neurologic, or cerebral disease (including demyelinating diseases such as multiple sclerosis) 25. Presence of a transplanted organ (with the exception of a corneal transplant > 3 months prior to screening) 26. Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence) 27. History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infra?clavicular, epitrochlear, or periaortic areas), or splenomegaly 28. Known recent substance abuse (drug or alcohol) 29. Poor tolerability of venipuncture or lack of adequate venous access for required blood sampling during the study period 30. Known atypical mycobacterium infection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2003-10; Study Completion 2005-12

PRIMARY OUTCOMES:
Fat-free mass

SECONDARY OUTCOMES:
Major Secondary Efficacy Endpoints in order of importance:
a. Change in body weight at 8 weeks
b. Change from baseline in functional capacity assessed by the incremental shuttle walk test (ISWT) at 8 weeks
c. Change from baseline in muscle strength (quadriceps, sniff nasal pressure, hand grip strength) at 8 weeks
d. Change from baseline in St George's Respiratory Disease Questionnaire (SGRQ) at 8 weeks
Other Secondary Efficacy Endpoints:
change from baseline at 8 weeks and other timepoints in:
a. Fat-Free Mass (FFM) as measured by DEXA scan
b. Body Mass Index (BMI)
c. Spirometry (FEV1, FVC, PEF25-75)
d. Quality of life as measured by the Short-Form 36-Item (SF-36)
e. Transitional Dyspnoea Index (TDI)
f. Muscle cell histology: muscle biopsy is optional
g. Sputum inflammatory cell count: sputum induction is optional
h. Exacerbation frequency and severity
Other objectives of this trial are to evaluate pharmacokinetics (PK) and pharmacodynamics (PD) in the treatment of patients with COPD-related cachexia.

CONTACTS AND LOCATIONS:
Overall Officials: Emiel FM Wouters, PhD, MD, Principal Investigator — University Hospital Maastricht, Department of Respiratory Medicine
Locations (1):
- Center for Integrated Rehabilitation and Organ failure (CIRO) Horn, Horn, Netherlands

REFERENCES:
- [Background] van der Vaart H, Koeter GH, Postma DS, Kauffman HF, ten Hacken NH. First study of infliximab treatment in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Aug 15;172(4):465-9. doi: 10.1164/rccm.200501-147OC. Epub 2005 Jun 3. PMID 15937294